CLINICAL TRIAL: NCT07188480
Title: The Role of DNA and RNA From Extracellular Vescicles Obtained by Bronchial Lavage in NGS Analyses for Advaced Stage NSCLC Patients
Brief Title: The Role of DNA and RNA in NGS Analyses for Advaced Stage NSCLC Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Gian Piero Bandelli, MD, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Geno_broncho_typing; RC24000851-2790626 (Other Grant/Funding Number: Ministero della Salute)
Record Dates: First submitted 2025-09-10; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Non Small Cell Lung Cancer NSCLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with suspected advanced lung cancer (Experimental): Patients with suspected advanced lung cancer undergo cytological and histological sampling via bronchoscopy, transthoracic or percutaneous procedures to confirm the diagnosis and, where deemed appropriate based on the characteristics of the cancer itself, to enable NGS analysis to be performed.
  Interventions: Diagnostic Test: bronchial lavage for NGS analysis

INTERVENTIONS:
Diagnostic Test: bronchial lavage for NGS analysis — NGS analysis conducted on bronchoscopic cytological samples in patients with NSCLC

SUMMARY:
Patients with advanced non-small cell lung cancer (NSCLC) usually undergo biopsies to obtain cytological material on which to perform Next Generation Sequencing (NGS) analysis, with the aim of identifying driver gene mutations that may be targeted by specific therapies. With the development of drugs with specific therapeutic targets, the clinical need for re-biopsy or even repeated biopsies is increasing; these biopsies are necessary to identify the mechanisms of drug resistance in the target lesions. Very often, lung cancer presents with small lesions and/or lesions located in areas that are difficult to reach with traditional biopsy techniques.

An alternative way to obtain genetic material is to isolate extracellular vesicles (EVs). These are secreted by almost all cell types, transport bioactive molecules, including nucleic acids (RNA and DNA), enclosed in a double lipid layer, and act as essential mediators in cell-cell communication. EVs are an ideal biomarker for cancer, as the content of EVs originating from tumor cells reflects the molecular and genetic composition of the parent cells. Long-stranded, concentrated EV-DNA is easy to amplify, making it a suitable candidate for NGS analysis. EVs are widely distributed in various body fluids, making them easier to sample using less invasive methods than tumor cells.

Recent studies have shown that EVs successfully isolated from bronchoalveolar lavage (BAL) fluid of lung cancer patients contain abundant amounts of dsDNA. In a study of patients with anatomopathologically confirmed NSCLC, the sensitivity and specificity of EGFR genotyping based on BAL EVs were high, and this test showed an even better mutation detection rate than tissue/cytology-based typing.

Considering the high positive predictive value of EV genotyping in bronchoalveolar lavage, this study aims to evaluate its feasibility in NGS analyses.

The primary objective of the study is to determine the technical feasibility of NGS analysis on EV-DNA/RNA derived from bronchoalveolar lavage in patients with advanced NSCLC.

The secondary objective is to determine the sensitivity and specificity of NGS analysis of EV-DNA/RNA derived from bronchoalveolar lavage compared to NGS analysis conducted on bronchoscopic cytological samples in patients with advanced NSCLC.

DETAILED DESCRIPTION:
In patients with advanced non-small cell lung cancer (NSCLC), who often undergo biopsies, there is a growing need to clearly define the clinical role of liquid biopsies. Lung tumors can only be visualized directly during bronchoscopy when located in central positions, sometimes making sampling difficult when they are located in more peripheral regions of the lung. With the development of drugs with specific therapeutic targets, the clinical need for re-biopsy or even repeated biopsies is increasing; these biopsies are necessary to identify the mechanisms of drug resistance in target lesions. Liquid biopsy of blood was introduced to overcome the difficulties in obtaining a quality solid tumor tissue sample through direct biopsy of tumor lesions, but it remains a secondary diagnostic technique compared to tissue biopsies due to its low sensitivity. Liquid biopsy of blood is a technique used to detect circulating deoxyribonucleic acid (DNA) derived from tumor cells (free DNA fragments in the blood). Furthermore, since blood is a complex body fluid consisting of many components, there is a need to identify a different biological resource from which to perform the liquid biopsy. In addition, the characteristics of 'naked' DNA ('Cell-Free DNA' - cfDNA) extracted from plasma after the removal of red blood cells have never been adequately defined, as this DNA may have originated from floating DNA, protein-DNA complexes and/or from within extracellular vesicles (EV). EVs, nano-sized vesicles secreted by almost all types of cells, transport bioactive molecules such as proteins, glycans, lipids, metabolites, and nucleic acids (RNA and DNA), enclosed in a double lipid layer, and act as essential mediators in cell-cell communication. EVs are an ideal biomarker for cancer, as the content of EVs originating from cancer cells reflects the molecular and genetic composition of the parent cells and is secreted in higher quantities than EVs from normal cells.

Researchers identified tumor-derived EVs carrying double-stranded DNA (dsDNA) and EV-DNA representing the entire genome, even reflecting the mutational status of the parental tumor cells. Several studies have also shown that, although EV-DNA exists in short and long sizes, most are 10 kb or longer, and have demonstrated that tumor-related mutations can be comprehensively detected using EV DNA. In addition, two types of DNA were identified, internally protected and external surface DNA, which could be used as a basis for the development of diagnostic methods.

Long-stranded, concentrated EV-DNA is easy to amplify, making it a suitable candidate for NGS analysis. It has been suggested that NGS analysis using EVs isolated from pleural effusion and urine could effectively replace NGS on tissue in cases where there is a shortage of tissue. The encapsulation of DNA within the double lipid layer of EVs appears to improve DNA stability by protecting it from the external environment. The amount of cfDNA released by tumors is normally low, representing only a fraction of the tumor's genomic heterogeneity released by dying tumor cells. In contrast, the process of isolating EVs from fluids increases the final concentration of EV-DNA obtained, and in addition, EVs are secreted by both viable and dying tumor cells. In a study comparing the use of EV-DNA and plasma cfDNA from NSCLC patients in liquid biopsies, EV-DNA improved the detection sensitivity of EGFR exon 19 deletion, L858R, and T790M mutations. This study also highlighted the diagnostic and prognostic capabilities of EV-DNA by demonstrating that mutations identifiable by liquid biopsy on EV-DNA included the specific acquired resistance mutation T790M. Furthermore, the specificity and sensitivity of liquid biopsy were further increased with the use of EV-DNA from bronchoalveolar lavage (BAL) fluid. EVs are widely distributed in various body fluids, making them easier to sample using less invasive methods than cancer cells. More importantly, specificity and sensitivity can increase significantly when EV-DNA is used for liquid biopsy compared to cfDNA. For these reasons, liquid biopsy using EV-DNA could be a clinically useful means of isolating cancer-specific DNA.

Lung cancer cells produce and release EVs in abundance in the tumor microenvironment (TME), which is easily accessible via bronchial wash (BW) or bronchoalveolar lavage (BAL). These procedures are mainly performed for diagnostic purposes, to obtain microbiological or cytological information from the main airways down to the subsegmental bronchi in the case of bronchial lavage, or from the lower respiratory tract and alveoli in the case of bronchoalveolar lavage. The results of liquid biopsy on EVs isolated from BAL and BW in patients with NSCLC have been shown to be superior to those of the same biopsy performed on plasma cfDNA. Recent studies have shown that EVs successfully isolated from BAL in patients with lung cancer contain abundant amounts of dsDNA, and that liquid biopsy for genotyping of the epidermal growth factor receptor (EGFR) using BAL is tissue-specific and extremely sensitive compared to the use of cfDNA. Furthermore, sensitivity increases proportionally with disease stage progression, reaching 100% in samples from stage IV patients. These results seem to suggest that EGFR genotyping from BAL-derived EVs is a highly promising liquid biopsy method, and particularly efficient for patients requiring repeated biopsies during disease progression. Furthermore, it is noteworthy that EGFR testing of BAL-derived EVs in stage I lung cancer showed a relatively high predictive value of 85.7%, despite a low sensitivity of 35.3%. BAL is a minimally invasive procedure associated with a low complication rate; however, it is technically more complex than bronchoalveolar lavage. The superiority of liquid biopsy was confirmed even on EV isolated from BW in patients with NSCLC compared to plasma cfDNA biopsy, achieving a diagnostic accuracy of 94.5% for EGFR genotyping.

In the diagnostic field, clinicians often find it difficult to manage slow-growing ground glass nodules (GGNs), especially in cases of low-intermediate risk of the lesion being tumorous. Three-quarters of resected GGNs tested positive for EGFR, KRAS, ALK, or HER2 mutations. Therefore, considering the high positive predictive value of EV genotyping on BAL and BW, the detection of a mutation through this sampling could be useful in directing treatment towards surgical resection rather than careful follow-up. The low sensitivity of the analysis could be improved by using more sensitive techniques such as next-generation sequencing and droplet digital PCR.

The results of this study will determine whether NGS analysis of EV-DNA/RNA (DNA/RNA derived from EVs) obtained from bronchial lavage is feasible in:

* patients with advanced-stage NSCLC for therapeutic purposes, avoiding more invasive forms of sampling;
* patients with GGN or lung tumors that cannot be sampled otherwise or can only be sampled surgically for diagnostic purposes.

This study is intended to be cross-sectional, feasibility-based, pilot, and experimental, exclusively on tissue samples. It will be conducted following prospective enrollment, in which each patient will undergo additional laboratory testing on a sample of fluid derived from bronchoalveolar lavage performed according to clinical practice.

In all patients with suspected advanced lung cancer requiring diagnostic confirmation by bronchoscopy, NGS analyses will be performed both on cytological samples taken by bronchoscopy (analysis performed according to clinical practice) and on EV-DNA/RNA derived from bronchial lavage (analysis covered by the study). In addition, in all patients with known NSCLC who have already undergone NGS analysis on cytological-histological samples, with an indication to perform a bronchoscopy for other reasons (microbiological or anatomical investigations), or in patients with known advanced-stage NSCLC who require cytological-histological retyping, including for NGS analysis in cases of suspected cancer progression, a subsequent NGS analysis will be performed on the EV-DNA/RNA (analysis covered by the study) on part of the bronchoalveolar lavage sample used for microbiological/cytological examination (clinical practice).

This study will enroll all adult patients, male and female, who have advanced-stage NSCLC requiring NGS analysis for therapeutic purposes, or who are indicated for bronchoalveolar lavage, having already undergone NGS analysis on cytological and histological samples in the previous five years.

In clinical practice, patients with suspected advanced lung cancer undergo cytological and histological sampling via bronchoscopy, transthoracic or percutaneous procedures to confirm the diagnosis and, where deemed appropriate based on the characteristics of the cancer itself, to perform NGS analysis.

In the patients under study, before performing any further cytological sampling by bronchoscopy with ancillary instruments (such as a needle or forceps), bronchial lavage will be performed at the site of interest, instilling saline solution as per normal clinical practice for cytological investigation.

The bronchial lavage fluid will be collected and subjected in part to cytological analysis as per normal clinical practice, and in part to EV isolation (subject of the study).

The isolation of EVs from bronchoalveolar lavage will be carried out by separation on a purification column following sequential centrifugation. The size distribution and number of extracellular vesicles will be analyzed using a laser nanoparticle characterization system called Nanoparticles Tracking Analysis (NTA), a tool available at the Transplant Immunobiology Laboratory. The analysis of the EV phenotype in BAL will be performed using two methods: flow cytometry and ExoView analysis. This analysis will allow the expression of characteristic EV protein markers such as CD63, CD9, and CD81 to be determined.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Indication for bronchoscopic cytological sampling for further diagnosis of suspected stage IV lung cancer on CT (computed tomography)/PET (positron emission tomography) scans, with consequent need for NGS analysis.
* Indication for bronchoscopy in patients with known lung cancer who have already undergone NGS analysis on a cytological-histological sample in the previous five years.
* Acquisition of written informed consent.

Exclusion Criteria:

* Confirmation of small cell lung cancer or other non-NSCLC pathology where there is no indication for NGS testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Adequacy ratio | Up to one year after the bronchoalveolar lavage
  Proportion of cases in which bronchoalveolar lavage allows sufficient and adequate material to be obtained for NGS analysis of EV-DNA/RNA, compared to the total number of patients undergoing bronchoalveolar lavage.

SECONDARY OUTCOMES:
Sensitivity and specificity of NGS analysis | Up to one month after the NGS analysis has been performed (up to one year after the bronchoalveolar lavage)
  To measure the sensitivity and specificity of NGS analysis on EV-DNA/RNA derived from bronchoalveolar lavage compared to NGS analysis conducted on bronchoscopic cytological samples, the genetic mutations obtained with the two methods will be compared, considering bronchoscopic cytological samples as a reference. NGS analyses will be performed for each patient enrolled in the study at the end of the bronchoscopic examination.

CONTACTS AND LOCATIONS:
Overall Officials: Gian Piero Bandelli, md, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy